CLINICAL TRIAL: NCT00263991
Title: Cortical Reorganisation in Patients With Primary Headache Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Danish Headache Center (Other)
Other Study IDs: KA 05085
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 2005-08

CONDITIONS: Migraine Without Aura; Chronic Tension-Type Headache
MeSH Terms: conditions — Migraine without Aura

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

INTERVENTIONS:
Device: EEC-techniques

SUMMARY:
Primary headache disorders are now accepted as physiological diseases, and advanced imaging-techniques have demonstrated a migraine generator in the brain stem and increased stimulus sensitivity in these patients. The underlying neuronal dysfunctions remain to to clarified and the existing neurophysiological methods have not yet been useful. More sensitive and reliable methods are therefore highly needed. The aims of the study are therefore to develop a sensitive and reliable method to demonstrate a cortical reorganisation and expansion of pain sensitive cortical areas in patients with migraine or tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis og migraine without aura or chronic tension-type headache

Exclusion Criteria:

* serious somatic or psychiatric diseases including depression
* overuse of analgesics
* regular intake of opiates or benzodiazepines
* intake of prophylactic headache medication
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bendtsen, MD, Ph.d, Principal Investigator — Danish Headache Center, Department of Neurology, Glostrup Hospital, University of Copenhagen, Denmark
Locations (1):
- Danish Headache Center; Department of Neurology, Glostrup Hospital, University of Copenhagen, Glostrup, Copenhagen, Denmark